CLINICAL TRIAL: NCT04648501
Title: The Role of Integrated Cognitive and Balance (Dual-task) Training in Balance and Fall Risk in Individuals With Cerebellar Ataxia: A Randomized Controlled Trial
Brief Title: Dual Task Training for Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); National University of Singapore (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0030895
Record Dates: First submitted 2020-11-11; First posted 2020-12-01 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2020-10

CONDITIONS: Cerebellar Ataxia
Keywords: Dual-task; Balance training; Fall prevention; Economic evaluation
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: An assessor and statistician blinded two-arm parallel group, RCT comparing dual-task (CIBT) to single-task (conventional balance, coordination and cognitive) training will be conducted with 44 participants with CA. Eligible participants will be randomized to study groups and allocation will be concealed. Participants will be randomized to one of the two groups: Group 1: Dual-task (CIBT) training; and Group 2: Single-task active control (conventional balance, coordination and cognition) training.
Who Masked: Outcomes Assessor
Masking Description: A person not involved in the study (student helper #1) will randomize participants to study groups in permuted blocks through computer-generated random numbers list prepared by The student helper who is not involved in the recruitment, assessment of study variables, or intervention delivery will perform the allocation of participants into the experimental group and active control groups. One other part-time research assistant will be recruited to conduct all the other methodological procedures of the project (RA2). Assessments will be performed by a PhD student of the PI who is blind to treatment condition. Statistical analysis will be performed by the PI who will be blind to treatment condition during analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task group (Experimental): Dual-task (CIBT- experimental) group participants will receive 10 minutes of warm up, 40 minutes of CIBT training and 10 minutes of cool down exercises. CIBT program includes performing four types of cognitive tasks during sit to stand, standing with feet apart, one leg, tandem standing, multidirectional reaching, stair climbing and walking (10 metres) tasks. The four cognitive tasks will include: counting backwards by subtracting 4 numbers (for mental tracking ), naming fruits, vegetables, or animals (for working memory), auditory cues for performing activities, example, perform heel raise when you hear the alphabet H (for improving attention and auditory discrimination), short story telling (for verbal fluency). In addition, falls prevention strategies will be taught.
  Interventions: Other: Dual-task training
- Single-task group (Active Comparator): Single-task (conventional balance, coordination and cognitive training- active control) group participants will receive 10 minutes of warm-up, 20 minutes of conventional balance and coordination exercises that are in accordance to previously published literature, 20 minutes of cognitive training as single-task (same 4 tasks provided for the CIBT) and 10 minutes of cool down. In addition, falls prevention strategies will also be taught.
  Interventions: Other: Dual-task training

INTERVENTIONS:
Other: Dual-task training — Dual-task (CIBT- experimental) group participants will receive 10 minutes of warm up, 40 minutes of CIBT training and 10 minutes of cool down exercises. CIBT program includes performing four types of cognitive tasks during sit to stand, standing with feet apart, one leg, tandem standing, multidirectional reaching, stair climbing and walking (10 metres) tasks. The four cognitive tasks will include: counting backwards by subtracting 4 numbers (for mental tracking ), naming fruits, vegetables, or animals (for working memory), auditory cues for performing activities, example, perform heel raise when you hear the alphabet H (for improving attention and auditory discrimination), short story telling (for verbal fluency). In addition, falls prevention strategies will be taught.
  Other Names: Physical and cognitive exercises

SUMMARY:
Combining cognitive training with physical training to improve balance is a new approach for reducing the risk of falls in patient populations who are at risk for falls. People with brain pathology including cerebellar ataxia (CA) have difficulty in performing dual-tasks. Deficiency in dual-task performance relative to single-task performance referred to as dual-task cost is high in CA. Due to the high demands on cognitive resources, people with CA have higher falls rates during activities that involve dual tasking. Tai-Chi involves both cognition and physical movements making it a dual-tasking activity. However, previous study on the effects of 12-weeks of 8-form Tai-Chi did not demonstrate that it had beneficial effects in reducing falls among CA population. This null finding could potentially be due to (1) the lower levels of cognitive demands of Tai-Chi exercise, (2) the intervention not being intensive enough, or (3) the intervention may not have targeted the specific symptoms of CA. To determine if adding structured cognitive demands to conventional balance and coordination training (i.e., addressing all three possibilities for our previous null findings), the investigaotrs conducted a pilot study (n=5) to evaluate the feasibility, safety and benefits of a Cognitive-coupled Intensive Balance Training (CIBT) program. The more intensive and focused CIBT intervention reduced dual-task cost, improved balance, and reduced the number of falls in a sample of individuals with CA. Important next steps is to (1) evaluate the efficacy of the CIBT in a fully powered clinical trial, (2) understand the mechanisms underlying the benefits of CIBT training, and (3) determine the cost-benefits of this intervention. The hypothesis for the study includes (1) CIBT will improve balance and reduce falls; (2) reduction in dual-task cost of balance and cognitive performance will mediate a reduction in the number of falls in CA and (3) CIBT will be a cost-effective treatment option for improving balance and reduce falls. To test these hypotheses, a randomized controlled trial (RCT) with economic evaluation will be conducted over a period of two years to evaluate the effectiveness and cost-effectiveness of dual-task (CIBT) training compared with single-task (conventional balance: active control) training in individuals with CA.

DETAILED DESCRIPTION:
Frequent falls in people with cerebellar ataxia (CA) is a significant problem because it increases the burden of disease to both the individual and the healthcare system. Therefore, an intervention that could improve balance and reduce the number of falls is of paramount importance from the patients' perspective. Although the incidence of CA in the population is not as high as the other neurological disorders such as stroke and Parkinson's disease, the disability and its negative impact on quality of life are significant for those suffering from CA. Moreover, research that results in more knowledge regarding the factors that contribute to falls and the efficacy of treatments that reduce falls in this population could inform research into fall prevention in other populations of individuals at risk for falls, including otherwise healthy elderly adults. Individuals with CA have poor coordination, balance and postural control; all of these contribute to them having frequent falls. People with CA also present with varying degrees of cognitive impairments making it difficult for them to perform dual-tasks in daily activities. Dual tasking has been found to deteriorate the performance of either or both tasks in people with CA. The deficiency in dual-task performance relative to single-task performance referred to as dual-task cost is high in CA. Falls incidence in people with CA increases during daily activities that involve dual tasking. Tai-Chi is a form of dual-task training. Previous study of the Tai-Chi to improve balance and prevent falls in people with CA found some beneficial effects of Tai-Chi on improving balance, but it did not reduce falls incidence. The investigaotrs speculate the lack of beneficial effects of Tai-Chi on falls incidence was due to the Tai-Chi intervention being inadequately intense, especially with respect to its cognitive demand. Other available interventions to improve balance and reduce falls do not address the dual-task cost of balance performance in this population. However, dual-task training is found to reduce dual-task cost and reduce falls in people other neurological disorders and therefore has the potential to reduce falls in CA. To evaluate this possibility, the investigators developed and piloted the Cognitive-coupled Intensive Balance Training (CIBT) that combines cognitive demand to intensive balance and coordination training for reducing the dual-task cost of balance and cognitive performance, improve balance and consequently reduce the number of falls. The pilot study found that CIBT is safe, feasible and potentially effective in reducing the dual-task cost of balance performance, improving functional balance and reducing falls in people with CA. Evaluating the efficacy of this program in a fully powered clinical trial and understanding the mechanisms underlying the effectiveness of the CIBT on balance and falls are important next steps of our research program. Here the investigators propose a randomized controlled trial (RCT) to compare the treatment benefits of the dual-task (experimental: CIBT) training against the single-task (active control: conventional balance, coordination and cognition) training for reducing dual-task cost, improving balance and reduce the number of falls in participants with CA, evaluating both the efficacy and the mechanisms of dual-task training. In addition, the investigators propose to conduct an economic evaluation alongside the RCT at a healthcare perspective of Hong Kong to compare the cost-effectiveness of dual-task training against single-task training, in preparation for the development of any future trials. This study finding will have important clinical implications by clarifying if adding a cognitive demand to routine balance and coordination training will result in additional benefits on improving balance and reducing falls in comparison with usual care in people with CA. The findings will also have important implications for increasing the efficacy of falls prevention programs in other populations with neurological deficits who are at risk for falls. Our specific objectives are:

Objective 1: To evaluate the effectiveness of the dual-task (CIBT- experimental) training compared with single task (conventional intensive balance, coordination and cognitive- active control) training on functional balance and number of falls.

Hypothesis 1: Both dual-task and single-task training will improve functional balance, however, the dual-task training will be more effective in reducing the number of falls.

Objective 2: To identify the mechanism underlying the effectiveness of the dual-task training on functional balance and the number of falls; that is, to evaluate the extent to which treatment-related changes in the functional balance and dual-task cost of balance and cognitive performance mediate the reduction in the number of falls.

Hypothesis 2: Improvement in functional balance resulting in the reduction of number of falls will be mediated by the reduction in the dual-task cost of balance and cognitive performances.

Objective 3: Compare the cost-effectiveness of the dual-task and single-task training for preventing falls.

Hypothesis 3: Dual-task training will be superior in terms of cost-effectiveness than the single-task from a health-care perspective of Hong Kong

ELIGIBILITY:
Inclusion Criteria:

* Men and women in the age group of 18-60 years;
* Confirmed diagnosis of CA (of any type);
* Able to walk independently with or without walking assistive aids.

Exclusion Criteria:

* Previous history of other neurological diseases (such as Parkinson's disease, stroke, or polyneuropathies) or musculoskeletal problems severely impairing balance, gait or motor performance;
* Able to walk only with handheld support
* Severe visual impairment preventing from exercise participation and
* Severe cognitive impairment with scores <16 on the Montreal Cognitive Assessment (MoCA) scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Dual-task cost of balance performance will be assessed for the TUG | 0 weeks
  Based on the scores of the standard TUG (single task), d-TUG (dual-task TUG) test and standard counting backwards, the dual-task cost of balance performance will be estimated using the formula: (d-TUG - Standard TUG)/ Standard-TUG) × 100.
Dual-task cost of balance performance will be assessed for the TUG | Change score at 10 weeks and 34 weeks
  Based on the scores of the standard TUG (single task), d-TUG (dual-task TUG) test and standard counting backwards, the dual-task cost of balance performance will be estimated using the formula: (d-TUG - Standard TUG)/ Standard-TUG) × 100.

SECONDARY OUTCOMES:
SOT | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Will be assessed using the Bertec ® system. Ability to stand unsupported in conditions challenging the visual, vestibular and somato-sensory inputs will be assessed.50 We will assess (1) equilibrium score using the center of gravity (COG) sway of each condition, (2) composite equilibrium score and (3) sensory analysis ratio.
Limits of stability (LOS) | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Will be assessed using the Bertec ® system. The LOS assesses the ability to shift weight in 8 difference directions. We will assess Reaction time (RT) and Maximal Excursion (MxE)
Number of falls | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Number of falls will be obtained used digital diary. We operationally define a fall as an event when the person ends up on the ground or other surfaces due to a trip or any other unintentional activity, and a near fall as an unexpected loss of balance that did not result in complete loss of upright standing.
Montreal Cognitive Assessment (MoCA), | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  MoCA estimates memory, executive function, attention, language, abstraction, naming, delayed recall and orientation.45 This brief tool scores cognitive function out of 30, with a higher score equating to better function.
Scale for the Assessment & Rating of Ataxia (SARA) | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Is a measure for rating severity of ataxia.52 SARA has eight sub-components with a total score of 40, higher scores indicating greater severity of symptoms due to ataxia. It is reported to have good reliability, validity and responsiveness in CA
Berg Balance Scale (BBS) | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Is a measure of dynamic balance scored out of 56, higher scores indicating better balance. The BBS is found reliable and validity in people with CA
EuroQol-5-dimension-5- level (EQ-5D-5L). | 0 weeks, 6 weeks, 10 weeks and 34 weeks
  Health status will be assessed using the EuroQol-5-dimension-5-level (EQ-5D-5L). It is a standardised measure of health status used for economic appraisal

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winser SJ, Chan AYY, Whitney SL, Chen CH, Pang MYC. Effectiveness and cost of integrated cognitive and balance training for balance and falls in cerebellar ataxia: a blinded two-arm parallel group RCT. Front Neurol. 2024 Jan 19;14:1267099. doi: 10.3389/fneur.2023.1267099. eCollection 2023. PMID 38313407